CLINICAL TRIAL: NCT02758314
Title: Clinical Pathological Features Associated With the Expression of PD1 / PD-L1 in Subpopulations of Peripheral Blood and Tumor Tissue in Patients With Advanced Non-small Cell Lung Cancer, Their Role as Prognostic and Therapeutic Targets
Brief Title: Evaluation of PD1 / PDL1 Expression on Blood Cells & Tumor Tissue, Their Role as a Prognostic Target in NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez MD, Director and Head of Functional Unit of Thoracic Oncology and Personalized Medicine Laboratory. SNI III, Instituto Nacional de Cancerologia de Mexico
Other Study IDs: INCAN/CI/498/13
Record Dates: First submitted 2016-04-06; First posted 2016-05-02 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: PD-1; PD-L1; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood cells, serum and plasma, tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases / NSCLC patients: Evaluation of PD-1/PDL-1 expression.
  Evaluate the expression of PD-1 / PD-L1 on T-cell subpopulations (CD3 + (CD4 +, CD8 +), B cells (CD19 + CD20 +), natural killer (NK) cells (CD16 + CD56 +) NK T-cells (CD3 + CD16 + CD56 + ) peripheral blood samples in 150 NSCLC, free treatment by flow cytometry.
  Evaluate the expression of PD-1 / PD-L1 in tumor tissue obtained by biopsy of patients with NSCLC by immunohistochemistry.
  The patients for the enrollment have to be diagnosed with advanced Non-Small Cell Lung Adenocarcinoma (clinical stages IIIA, IIIB and IV), treated at the Instituto Nacional de Cancerología (INCan) who had not received radiotherapy and / or chemotherapy prior to obtaining samples to analyze. ECOG performance status 0-2 and present evidence of measurable disease.
  Interventions: Other: Evaluation of PD-1/PDL-1 expression.
- Control / Healthy subjects: Evaluation of PD-1/PDL-1 expression.
  Evaluate the expression of PD-1 / PD-L1 on T-cell subpopulations (CD3 + (CD4 +, CD8 +), B cells (CD19 + CD20 +), natural killer (NK) cells (CD16 + CD56 +) NK T-cells (CD3 + CD16 + CD56 + ) peripheral blood samples in 50 samples, by flow cytometry.
  Healthy subjects blood cells will be obtained from the blood bank at the Instituto Nacional de Cancerología (INCan)
  Interventions: Other: Evaluation of PD-1/PDL-1 expression.

INTERVENTIONS:
Other: Evaluation of PD-1/PDL-1 expression. — Evaluate the expression of PD-1 / PD-L1 on T-cell subpopulations of peripheral blood by flow cytometry and in tumor tissue by immunohistochemistry in NSCLC, free treatment and healthy subjects

SUMMARY:
Several reports have examined Programmed Death 1 (PD-1) expression on tumor-infiltrating T-cells, and its correlation with prognosis has been discussed. However, Programmed Death 1 (PD1)/Programmed Death Ligand 1 (PDL1) expression on the peripheral blood T-cells of cancer patients, particularly in those with lung cancer, has not been sufficiently studied. The purpose of this study is evaluate the expression of PD1 and PDL1 in subpopulations of peripheral blood and tumor cells patients with lung cancer non-small cell (NSCLC), associating with clinicopathological features of the patients studied.

DETAILED DESCRIPTION:
This is a prospective cohort study including patients with NSCLC stages IIIA, IIIB and IV lung cancer clinic of the National Cancer Institute (INCAN)

Clinical samples. Prior and informed consent before receiving any treatment, sample be obtained 15 ml peripheral blood of each subject included in the study (patients and controls). mononuclear peripheral blood cells (PBMC) from different groups of subjects separated by centrifugation gradient (Polymorphprep, Accurate Chemical) are used. The cells are resuspended in dimethylsulfoxide (DMSO) and 10% fetal bovine serum (FBS) to 90% at a concentration of 1 million cells per ml and kept in liquid nitrogen until use.

Evaluation of PD-1, PD-L1 by flow cytometry. The following monoclonal antibodies directed against cell surface antigens of human are used: anti-PD-1, anti-PD-L1, anti-PD-L2, anti- cluster of differentiation (CD) 3, anti-CD4, anti-CD8, anti-CD14, anti-CD16, anti-CD56, anti-CD19, anti-CD20.

Immunolocalization of PD-1, PD-L1 in lung tumor tissue of patients with NSCLC. Immunohistochemical staining (IHC). Lung biopsy is obtained paraffin blocks, and are processed by IHC technique for antitumor expression of PD1 / PDL1.V PD-L1 immunostaining was classified into two groups according to intensity and extent: (a) negative, when no staining or positive staining was detected in <5% of the cells; and (b) positive, when membranous staining was present in P5% of the cells.

ELIGIBILITY:
Inclusion Criteria patient :

1. Patients who have understood and signed the informed consent.
2. Diagnosis of lung cancer, histologically or cytologically documented (stage IIIA / B or IV) non-small cell adenocarcinoma, which had not received radiotherapy and / or chemotherapy prior to the first sample.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 and evidence of measurable disease.

Exclusion Criteria patient:

1. Subjects with Non-small cell lung cancer with a different histological type to adenocarcinoma.
2. Subjects with acute inflammation and uncontrolled infections.

Inclusion Criteria healthy subjects :

1. Informed consent in writing (signed) to participate in the study.
2. No diagnosis of oncological disease.
3. Subjects without symptoms of any respiratory illness in the two weeks prior to sampling.

Exclusion criteria healthy volunteers.

1. Any unstable systemic disease (including active or metabolic infection, congestive heart failure, liver disease, kidney).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It will include patients diagnosed with advanced non-small cell lung adenocarcinoma (clinical stages IIIA, IIIB and IV) treated at the Instituto Nacional de Cancerología (INCan).
  Subjects without previous radiotherapy and / or chemotherapy (prior sampling).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Immunolocalization of PD-1, PD-L1 in lung tumor tissue of patients with NSCLC. Immunohistochemical staining (IHC) | Baseline evaluation
  Immunolocalization of PD-1, PD-L1 in lung tumor tissue of patients with NSCLC. Immunohistochemical staining (IHC). Lung biopsy is obtained paraffin blocks, and are processed by IHC technique for antitumor expression of PD1 / PDL1.V PD-L1 immunostaining was classified into two groups according to intensity and extent: (a) negative, when no staining or positive staining was detected in <5% of the cells; and (b) positive, when membranous staining was present in P5% of the cells.

SECONDARY OUTCOMES:
Evaluation of PD-1, PD-L1 by flow cytometry. | Baseline evaluation
  Evaluation of PD-1, PD-L1 by flow cytometry. The following monoclonal antibodies directed against cell surface antigens of human are used: anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cluster of differentiation 3 (CD3), anti-CD4, anti-CD8, anti-CD14, anti-CD16, anti-CD56, anti-CD19, anti-CD20.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Gerardo MD Arrieta Rodriguez, Oncology, Principal Investigator — Instituto Nacional de Cancerologia, Mexico
Locations (1):
- Instituto National de Cancerologia, México, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gajewski TF, Schreiber H, Fu YX. Innate and adaptive immune cells in the tumor microenvironment. Nat Immunol. 2013 Oct;14(10):1014-22. doi: 10.1038/ni.2703. PMID 24048123
- [Background] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Background] Pennock GK, Chow LQ. The Evolving Role of Immune Checkpoint Inhibitors in Cancer Treatment. Oncologist. 2015 Jul;20(7):812-22. doi: 10.1634/theoncologist.2014-0422. Epub 2015 Jun 11. PMID 26069281
- [Background] Su M, Huang CX, Dai AP. Immune Checkpoint Inhibitors: Therapeutic Tools for Breast Cancer. Asian Pac J Cancer Prev. 2016;17(3):905-10. doi: 10.7314/apjcp.2016.17.3.905. PMID 27039716
- [Derived] Arrieta O, Montes-Servin E, Hernandez-Martinez JM, Cardona AF, Casas-Ruiz E, Crispin JC, Motola D, Flores-Estrada D, Barrera L. Expression of PD-1/PD-L1 and PD-L2 in peripheral T-cells from non-small cell lung cancer patients. Oncotarget. 2017 Oct 24;8(60):101994-102005. doi: 10.18632/oncotarget.22025. eCollection 2017 Nov 24. PMID 29254220